CLINICAL TRIAL: NCT01516671
Title: Pilot Study on the Role of Neuroinflammation in the Pathophysiology of Subarachnoid Hemorrhage and the Value of the Bilateral Bispectral Index for Early Diagnosis of Cerebral Ischemia After Subarachnoid Hemorrhage.
Brief Title: Neuroinflammation and Bispectral Index After Subarachnoid Hemorrhage
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Cyrill Hornuss, Study Principal Investigator, Ludwig-Maximilians - University of Munich
Other Study IDs: LMU-XX2011
Record Dates: First submitted 2012-01-16; First posted 2012-01-25 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Subarachnoid Hemorrhage
Keywords: Subarachnoid hemorrhage; Cerebral vasospasm; Neuroinflammation; Bilateral Bispectral Index
MeSH Terms: conditions — Subarachnoid Hemorrhage; Vasospasm, Intracranial; Neuroinflammatory Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cerebrospinal fluid Blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Subarachnoid hemorrhage (SAH) is associated with a high mortality and frequently leads to severe disability in survivors caused by cerebral vasospasm and infarction.

This study aims to elucidate the role of neuroinflammation (endocannabinoids and cortisol levels in cerebrospinal fluid) in the pathophysiology of cerebral vasospasm and the value of the bilateral bispectral index (BIS) for the early diagnosis of cerebral vasospasm.

DETAILED DESCRIPTION:
Subarachnoid hemorrhage (SAH) or bleeding in the brain is a form of stroke. SAH mostly results from ruptured aneurysms. This severe disease often results in death or severe physical or cognitive disabilities and reduced quality of life. One frequent complication after SAH is cerebral vasospasm, a spasm of the big arteries accompanied by infarction of healthy brain tissue. The pathophysiologic processes which drive vasospasm remain unclear. This study aims to examine the role of endocannabinoids and cortisol in cerebrospinal fluid during the development of cerebral vasospasm. Additionally, this study examines whether side difference in the processed electroencephalogram (bilateral bispectral index) may be useful for early detection of cerebral vasospasm.

ELIGIBILITY:
Inclusion Criteria:

* Admission to neurosurgical ICU Klinikum der Universität München
* SAH
* External CSF drainage

Exclusion Criteria:

- AGE < 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after acute SAH admitted to neurosurgical ICU
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Concentrations of endocannabinoids and corticoids in cerebrospinal fluid and blood. | Once per day from day 1 until day 14 after hospital admission
  Samples of cerebrospinal fluid and blood will be collected every day at 8am on hospital day 1-14 and the concentrations of the following substances will be determined:
  1. Anandamide
  2. 2-arachidonoylglycerol
  3. 2-arachidonoylglycerol-ether
  4. N-arachidonoyldopamine
  5. N-arachidonylglycine
  6. O-arachidonylethanolamide
  7. Palmitoylethanolamide
  8. Cortisol
  9. Corticotropin-releasing hormone (in CSF only)
  10. Corticosteroid-binding globulin (in blood only)
Bilateral Bispectral Index | Every second from 0:01 am until 23:59 pm on hospital day 1,2,3,4,5,6,7,8,9,10,11,12,13,14
  The Bispectral Index is calculated every second by the BIS Vista monitor. These data will be recorded continuously from 0:01 am until 23:59 pm.

SECONDARY OUTCOMES:
Transcranial Doppler | Every day at 8 am from day 1 until day 14 after hospital admission
  The mean velocities in middle cerebral and anterior cerebral arteries will be determined by transcranial Doppler

CONTACTS AND LOCATIONS:
Overall Officials: Volker Huge, MD, Principal Investigator — Klinikum der Universität München, Ludwig-Maximilians-University, Department of Anaesthesiology; Cyrill Hornuss, MD, Principal Investigator — Klinikum der Universität München, Ludwig-Maximilians-University, Department of Anaesthesiology
Locations (1):
- Klinikum der Universität München, München, Germany

REFERENCES:
- [Background] Altay T, Smithason S, Volokh N, Rasmussen PA, Ransohoff RM, Provencio JJ. A novel method for subarachnoid hemorrhage to induce vasospasm in mice. J Neurosci Methods. 2009 Oct 15;183(2):136-40. doi: 10.1016/j.jneumeth.2009.06.027. Epub 2009 Jul 1. PMID 19576247
- [Background] Huge V, Lauchart M, Magerl W, Beyer A, Moehnle P, Kaufhold W, Schelling G, Azad SC. Complex interaction of sensory and motor signs and symptoms in chronic CRPS. PLoS One. 2011 Apr 29;6(4):e18775. doi: 10.1371/journal.pone.0018775. PMID 21559525
- [Background] Huge V, Lauchart M, Forderreuther S, Kaufhold W, Valet M, Azad SC, Beyer A, Magerl W. Interaction of hyperalgesia and sensory loss in complex regional pain syndrome type I (CRPS I). PLoS One. 2008 Jul 23;3(7):e2742. doi: 10.1371/journal.pone.0002742. PMID 18648647
- [Background] Provencio JJ, Altay T, Smithason S, Moore SK, Ransohoff RM. Depletion of Ly6G/C(+) cells ameliorates delayed cerebral vasospasm in subarachnoid hemorrhage. J Neuroimmunol. 2011 Mar;232(1-2):94-100. doi: 10.1016/j.jneuroim.2010.10.016. Epub 2010 Nov 6. PMID 21059474
- [Background] Lin CL, Dumont AS, Calisaneller T, Kwan AL, Hwong SL, Lee KS. Monoclonal antibody against E selectin attenuates subarachnoid hemorrhage-induced cerebral vasospasm. Surg Neurol. 2005 Sep;64(3):201-5; discussion 205-6. doi: 10.1016/j.surneu.2005.04.038. PMID 16099244
- [Background] Wolf SA, Tauber S, Ullrich O. CNS immune surveillance and neuroinflammation: endocannabinoids keep control. Curr Pharm Des. 2008;14(23):2266-78. doi: 10.2174/138161208785740090. PMID 18781977
- [Background] Tischner D, Reichardt HM. Glucocorticoids in the control of neuroinflammation. Mol Cell Endocrinol. 2007 Sep 15;275(1-2):62-70. doi: 10.1016/j.mce.2007.03.007. Epub 2007 May 4. PMID 17555867
- [Background] Annane D, Bellissant E, Bollaert PE, Briegel J, Confalonieri M, De Gaudio R, Keh D, Kupfer Y, Oppert M, Meduri GU. Corticosteroids in the treatment of severe sepsis and septic shock in adults: a systematic review. JAMA. 2009 Jun 10;301(22):2362-75. doi: 10.1001/jama.2009.815. PMID 19509383